CLINICAL TRIAL: NCT02424253
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Determine the Effects of 8 Weeks Treatment With Oral ZPL-3893787 (30 mg od x 56 Days) on Pruritus in Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Determine the Efficacy of ZPL-3893787 in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ziarco Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZPL389/101
Record Dates: First submitted 2015-04-17; First posted 2015-04-23 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZPL-3893787 (Experimental): 30 mg ZPL-3893787 orally once daily for 8 weeks.
  Interventions: Drug: ZPL-3893787
- Placebo (Placebo Comparator): 1 capsule orally once daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZPL-3893787 — ZPL-3893787
  Arms: ZPL-3893787
Drug: Placebo — Matched Placebo
  Arms: Placebo

SUMMARY:
This was a randomized, double blind, placebo controlled, parallel group study in approximately 90 subjects with moderate-severe AD Eczema Area and Severity Index (EASI) ≥12 and ≤ 48 (0-72 scale). Following a run-in subjects were randomized to receive either oral 30 mg ZPL-3893787 once daily (od) or placebo od for 8 weeks (56 days).

ELIGIBILITY:
Inclusion Criteria:

Males and females aged 18-65 years inclusive with physician documented history or diagnosis of atopic dermatitis for at least 12 months prior to screening. Chronic AD should be diagnosed by the Eichenfield revised criteria of Hanifin and Rajka (Eichenfield, 2004)

Eczema Area and Severity Index (EASI) of ≥12 and <48.

An Investigator's Global Assessment (IGA) score ≥ 3 at both Screening and Day 0.

A mean pruritus score of ≥ 5 on a 0-10 scale over the 7 day Run In (Days -7 to -1)

Atopic dermatitis affecting ≥10% BSA

Exclusion Criteria:

AD of such severity (EASI >48) that the subject could not comply with the demands of the study and/or the subject is not a suitable candidate for a placebo-controlled study

Have concurrent skin disease (e.g. acne) of such severity in the study area that it could interfere with the study evaluation or presence of skin comorbidities that may interfere with study assessments.

Have an active skin infection or any other clinically apparent infections.

Hypersensitivity to mometasone or to any other ingredients contained by the topical corticosteroid product used as rescue medication in the study.

Have received phototherapy (e.g. UVA, UVB), or systemic therapy (e.g. immunosuppressants, cytostatics) known or suspected to have an effect on AD, within 4 weeks of the start of the Run In.

Have received systemic corticosteroids ([CS] e.g. oral, intravenous, intraarticular, rectal) within 4 weeks of the start of the Run in. Subjects on a stable maintenance dose (over the preceding 3 months) of inhaled or intranasal CS may participate.

Were treated with oral antihistamines or topical calcineurin inhibitors or topical steroids within 7 days of starting Run In; intranasal antihistamines for the treatment of allergic rhinitis are acceptable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals
Locations (17):
- Belgium (3):
  - Belgium Study Site, Brussels
  - Belgium Study Site, Leuven
  - Belgium Study Site, Liège
- Germany (5):
  - German Study Site, Goch
  - German Study Site, Hamburg
  - German Study Site, Hanover
  - German Study Site, Mainz
  - German Study Site, Münster
- Poland (5):
  - Polish Study Site, Bialystok
  - Polish Study Site, Gdansk
  - Polish Study Site, Lodz
  - Polish Study Site, Poznan
  - Polish Study Site, Tarnów
- United Kingdom (4):
  - UK Study Centre, Blackpool
  - UK Study Centre, Cannock
  - UK Study Centre, Leeds
  - UK Study Centre, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first informed consent was on 18 May 2015. Subjects were randomly assigned 2:1 to receive either 30 mg ZPL-3893787 or matching placebo. The randomization was stratified by baseline worst daily pruritus NRS score (≤ 7.5 and > 7.5) determined from the mean pruritus score (worst itch over 24 hours) collected during the 7-day Run-in Period.
Period: Overall Study
Arm/Group | ZPL-3893787 | Placebo
Started | 65 | 33
Completed | 54 | 24
Not Completed | 11 | 9
Not completed — Other, unspecified | 1 | 0
Not completed — Compliance problems | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Lack of Efficacy | 0 | 7
Not completed — Adverse Event | 2 | 0
Not completed — Consent withdrawn by subject | 4 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): Included all randomized subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | ZPL-3893787 | Placebo | Total
Number analyzed (Participants) | 65 | 33 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (11.22) | 35.5 (12.52) | 34.3 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 20 | 56
  Male | 29 | 13 | 42
Fitzpatrick Skin Type [Number; unit: participants] — The Fitzpatrick scale is a numerical classification schema for human skin color. The scale ranges from I to VI and is defined as:
  Type I - always burns, never tans (palest; freckles). Type II - usually burns, tans minimally Type III - sometimes mild burn, tans uniformly Type IV - burns minimally, always tans well (moderate brown) Type V - very rarely burns, tans very easily (dark brown) Type VI - never burns (deeply pigmented dark brown to darkest brown)
  participants
    Type I | 2 | 4 | 6
    Type II | 24 | 11 | 35
    Type III | 32 | 14 | 46
    Type IV | 3 | 2 | 5
    Type V | 3 | 1 | 4
    Type VI | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Numerical Rating Score (NRS) for Pruritus (Worst Itch)
Description: The participant used the Pruritus NRS to rate his or her worst itch in the previous 12 hours. This was assessed twice daily (in the morning soon after rising and the evening prior to retiring) and recorded in the eDiary. The scale ranges from 0 (no itching) to 10 (itching as bad as can be imagined).
  If only 1 measurement was collected on a particular day, that score was counted as the worst measurement.
Time Frame: Baseline to Week 8
Population: Full Analysis Set (FAS): Included all randomized subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ZPL-3893787 | Placebo
Number analyzed (Participants) | 65 | 33
score on a scale
  Baseline summary | 7.3 (1.139) | 7.26 (1.054)
  Week 8 summary | 4.27 (2.253) | 4.6 (1.95)
  Change from Baseline | -3.03 (2.186) | -2.66 (2.057)
Statistical Analysis 1: Comparison: ZPL-3893787 vs Placebo; Change from baseline; Test type: Superiority; p = 0.249, ANCOVA — 1-sided p-value; The ANCOVA model included baseline value and treatment; LS Difference = -0.35, 90% CI 2-sided [-1.21 to 0.51]

2. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: The EASI is a validated tool used to measure the severity and extent of atopic eczema over 4 body regions (head and neck, upper limbs, trunk, and lower limbs). The intensity of a representative area of eczema and the approximate percentage affected by eczema are calculated for each region. A representative area of eczema is selected for each body region. The intensity of redness (erythema), thickness (induration, papulation, and edema), scratching (excoriation), and lichenification (lined skin) of eczema is assessed as:
  0 - None
  1. - Mild
  2. - Moderate
  3. - Severe The total score incorporates the extent of body regions affected. Scores range from 0 to 72 with higher scores indicating more severe eczema.
  Total score is calculated by summing the EASI scores of 6 symptoms across 4 body regions
Time Frame: Baseline to Week 8
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ZPL-3893787 | Placebo
Number analyzed (Participants) | 65 | 33
score on a scale
  Baseline | 21.39 (7.889) | 20.44 (6.868)
  Week 8 summary | 10.67 (9.541) | 15.06 (11.159)
  Week 8 change from baseline | -10.72 (9.679) | -5.38 (9.922)
Statistical Analysis 1: Comparison: ZPL-3893787; Change from baseline analysis; Test type: Superiority; p = 0.01, ANCOVA — 1-sided p-value; The ANCOVA model included baseline EASI, stratification variable (worst daily pruritus NRS ≤ 7.5 or > 7.5) and treatment; LS Difference = -5.06, 90% CI 2-sided [-8.66 to -1.46]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Screening to up to 28 days post last dose, up to approximately 10 months.
Arm/Group | ZPL-3893787 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/65 | 1/33
Other Adverse Events (participants affected / at risk) | 15/65 | 10/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZPL-3893787 (N=65) | Placebo (N=33)
Ulcerative keratitis (ulcus corneae left eye) (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZPL-3893787 (N=65) | Placebo (N=33)
Bradycardia (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 4
Somnolence (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Drug ineffective (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Decreased activity (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of the agreements with investigators may vary. However, the investigator is not prohibited from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.